CLINICAL TRIAL: NCT01606176
Title: A Multi Centre Randomised, Double Blind, Placebo Controlled, Parallel Group Comparison of the Effects of Cannabis Based Medicine Standardised Extracts Over 4 Weeks, in Patients With Chronic Refractory Pain Due to Multiple Sclerosis or Other Defects of Neurological Function.
Brief Title: A Study to Evaluate the Effects of Cannabis Based Medicine in Patients With Pain of Neurological Origin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWPS0105
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Pain; Multiple Sclerosis
MeSH Terms: conditions — Pain; Multiple Sclerosis | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GW-1000-02 (Experimental): Each 100 μl actuation contains 2.5 mg delta-9-tetrahydrocannabinol (THC) and 2.5 mg cannabidiol (CBD). The maximum permitted dose was 48 actuations in any 24 hour period (120 mg THC/120 mg CBD).
  Interventions: Drug: GW-1000-02
- Placebo (Placebo Comparator): Each 100 μl actuation contains the excipients only. The maximum permitted dose was 48 actuations in any 24 hour period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW-1000-02 — Each actuation of GW-1000-02 (100 μl) delivered a dose containing 2.5 mg delta-9-tetrahydrocannabinol (THC) and 2.5 mg cannabidiol (CBD). The maximum permitted dose of study medication was eight actuations in any three hour period (20 mg THC/20 mg CBD) and 48 actuations in any 24 hour period (120 mg THC/120 mg CBD).
  Other Names: Sativex
  Arms: GW-1000-02
Drug: Placebo — Each actuation of placebo (100 μl) delivered the excipients only. The maximum permitted dose of study medication was eight actuations in any three hour period and 48 actuations in any 24 hour period.
  Arms: Placebo

SUMMARY:
To investigate the ability of a cannabis based medicine extract to relieve chronic refractory pain of neurological origin.

DETAILED DESCRIPTION:
Patients with Multiple Sclerosis or other defect of neurological function with a qualifying symptom of chronic refractory pain, entered a seven day baseline period, followed by a 21 day randomised, double blind, parallel group comparison of GW-1000-02 with placebo, self-titrated to symptom resolution or maximum tolerated dose. The ability of the cannabis based medicine extract to relieve chronic refractory pain was assessed by the change from baseline in pain score using Box Scale-11 (BS-11) scores recorded in the patients' daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Patient, or legal representative, willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with chronic refractory pain due to Multiple Sclerosis or other defects of neurological function.
* Diagnosed with pain, not wholly alleviated with current analgesic therapy at Visit 1 and an average score of over 4 on a Box Scale-11 scale on the four consecutive days leading up to Visit 2, where: zero = "no pain" and 10 = "worst possible pain".
* Stable dose of pain relieving medication for at least two weeks prior to study entry.
* Willing to ensure that they or their partner use effective contraception during the study and for three months thereafter (applicable to female patients of child bearing potential and male patients whose partners were of child bearing potential).
* No cannabinoid use (cannabis, Marinol or Nabilone) for at least seven days before Visit 1 and be willing to abstain from any use of cannabis during the study.
* Able (in the investigator's opinion) and willing to comply with all study requirements.
* Willing for his or her name to be notified to the Home Office for participation in this study.
* Willing to allow his or her general practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* History of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* Known history of alcohol or substance abuse.
* Severe cardiovascular disorder, such as ischaemic heart disease, arrhythmias (other than well controlled atrial fibrillation), poorly controlled hypertension or severe heart failure.
* History of epilepsy.
* Female patients who were pregnant, lactating or planning pregnancy during the course of the study.
* Significant renal or hepatic impairment.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Terminally ill or inappropriate for placebo medication.
* Any other significant disease or disorder which, in the opinion of the investigator, may have put the patient at risk because of participation in the study, or may have influenced the result of the study, or the patient's ability to participate in the study.
* Regular levodopa (Sinemet®, Sinemet Plus®, Levodopa, L-dopa, Madopar®, Benserazide) therapy within seven days of study entry.
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medications.
* Known or suspected of having adverse reaction to cannabinoids.
* Travel outside the UK planned during the study.
* Donation of blood during the study.
* Patients who had participated in another research study in the 12 weeks leading up to study entry.
* Patients who had been previously randomised into this study.
* Male patients who were receiving Sildenafil (Viagra®) at the time of study entry and were unwilling to stop medication for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-03; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- James Paget Hospital, Norfolk, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- GW-1000-02: Each actuation of oromucosal spray delivers 2.5mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). The maximum permitted dose of was eight actuations in any three hour period, and 48 actuations in any 24 hour period (THC 120 mg : CBD 120 mg).
- Placebo: Placebo control. The maximum permitted dose of was eight actuations in any three hour period, and 48 actuations in any 24 hour period.
Period: Overall Study
Arm/Group | GW-1000-02 | Placebo
Started | 36 | 34
Completed | 32 | 31
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Disease progression | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GW-1000-02: Active treatment.
- Placebo: Placebo control.
- Total: Total of all reporting groups
Arm/Group | GW-1000-02 | Placebo | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 26 | 56
  >=65 years | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.72 (12.11) | 57.61 (10.28) | 54.58 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 16 | 13 | 29
Region of Enrollment [Number; unit: participants]
  United Kingdom | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Pain Box Scale-11 Score at 3 Weeks.
Description: Each day, in the morning (on waking), at lunchtime and in the evening (just before going to bed), patients recorded in their patient diary their level of pain using a Box Scale-11 pain score ranging from zero "no pain" to 10 "worst possible pain". Week 3 analysis was defined as the mean of the last seven days in the study. The last day was taken as the last day with complete diary card pain data that occurred on or before the last day the patient took study medication. A negative value from baseline indicates and improvement.
Time Frame: 0 - 3 weeks
Population: All patients who were randomised, received at least one actuation of study medication and completed at least one set of efficacy assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- GW-1000-02: Each 100 ul actuation contains 25 mg THC and 25 mg CBD. A maximum of 48 actuations (120 mg each of THC and CBD) was permitted in any 24 hour period.
- Placebo: Each 100 ul actuation contains the excipients. A maximum of 48 actuations was permitted in any 24 hour period.
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 36 | 34
units on a scale | -1.3 (1.67) | -0.9 (1.62)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change was compared between treatment groups using analysis of covariance (ANCOVA). The significance of the treatment effect, after adjusting for baseline pain score, was assessed using the F-test from the ANCOVA. The model was as follows: Change in Box Scale-11 Pain Score = Baseline Pain Score + Treatment; Test type: Superiority or Other; p = 0.332, ANCOVA; Estimated mean treatment difference = -0.39, 95% CI 2-sided [-1.18 to 0.40]

2. Secondary Outcome: Use of Analgesic Escape Medication.
Description: The percentage of days on treatment on which escape medication was used is presented.
Time Frame: 0 - 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 36 | 34
percentage of days | 20.57 (33.08) | 50.12 (44.10)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The proportions were compared between treatment groups using analysis of variance (ANOVA) with treatment as a factor; Test type: Superiority or Other; p = 0.002, ANOVA; Estimated mean treatment difference = -29.55, 95% CI 2-sided [-48.08 to -11.02]

3. Secondary Outcome: Change From Baseline in Mean Sleep Disturbance Score at 3 Weeks.
Description: Each day patients were asked to record in their patient diary, whether or not they were woken due to pain the previous night. Answers were recorded as "No", "Once", "Twice", "More than twice" and "Awake most of the night"; these were converted to a five point scale, zero to four, respectively. Sleep disturbance was summarised and analysed in the same manner as the analysis of the primary efficacy parameter of Box Scale-11 pain score. A negative value from baseline indicates and improvement.
Time Frame: 0 - 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 36 | 34
units on a scale | -0.57 (0.85) | -0.34 (0.58)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change was compared between treatment groups using ANCOVA. The significance of the treatment effect, after adjusting for baseline sleep disturbance score, was assessed using the F-test from the ANCOVA. The model was as follows: Change in Sleep Disturbance Score = Baseline Sleep Disturbance Score + Treatment; Test type: Superiority or Other; p = 0.052, ANCOVA; Estimated mean treatment difference = -0.34, 95% CI 2-sided [-0.68 to 0.00]

4. Secondary Outcome: Change From Baseline in Mean Total Pain Disability Index Score at 3 Weeks.
Description: The index consists of seven assessments of pain (representing different aspects) with each assessment scored on a zero "no disability" to 10 "total disability" scale. The total Pain Disability Index was calculated as the un-weighted sum of the seven pain scores; if one or more of the pain scores were missing then the total Pain Disability Index was set to missing. A reduction in score from baseline indicates and improvement.
Time Frame: 0 - 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 28 | 26
units on a scale | -5.9 (10.17) | -3.2 (9.77)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change was compared between treatment groups using ANCOVA. The significance of the treatment effect, after adjusting for baseline Pain Disability Index score, was assessed using the F-test from the ANCOVA. The model was as follows: Change in Pain Disability Index Score = Baseline Pain Disability Index Score + Treatment; Test type: Superiority or Other; p = 0.300, ANCOVA; Mean Difference (Final Values) = -2.79, 95% CI 2-sided [-8.14 to 2.56]

5. Secondary Outcome: Change From Baseline in Mean Total Brief Pain Inventory (Short Form) Score at 3 Weeks.
Description: The Brief Pain Inventory (Short Form) is a 14-item questionnaire that asks patients to rate pain over the prior week and the degree to which it interferes with activities on a 0 to 10 scale, where 0=no pain and 10=pain as bad as you can imagine. Severity is measured as worst pain, least pain, average pain, and pain right now. The severity composite score was calculated as the arithmetic mean of the four severity items (range 0-10). The minimum value is zero and maximum is 10. A reduction in score from baseline indicates an improvement.
Time Frame: 0 - 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 34 | 34
units on a scale | -3.6 (5.12) | -1.9 (6.52)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change was compared between treatment groups using ANCOVA. The significance of the treatment effect, after adjusting for baseline Total Brief Pain Inventory (Short Form) score, was assessed using the F-test from the ANCOVA. The model was as follows: Change in Total Brief Pain Inventory (Short Form) Score = Baseline Total Brief Pain Inventory (Short Form) Score + Treatment; Test type: Superiority or Other; p = 0.233, ANCOVA; Estimated mean treatment difference = -1.66, 95% CI 2-sided [-4.42 to 1.10]

6. Secondary Outcome: Change From Baseline in Mean Spitzer Quality of Life Index Scores at 3 Weeks.
Description: The Spitzer Quality of Life Index questionnaire consists of five sections, relating to activity, daily living, health, support and outlook. Each section has three choices (numbered 1, 2 and 3) and the patient was required to choose the one that best described their quality of life during the last week. Choice 1 is scored two, Choice 2 is scored one and Choice 3 is scored zero. The total Spitzer Quality of Life Index was calculated as the unweighted sum of the five scores. A reduction in score from baseline indicates an improvement.
Time Frame: 0 - 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 33 | 31
units on a scale | -0.2 (1.17) | -0.4 (1.54)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The change was compared between treatment groups using ANCOVA. The significance of the treatment effect, after adjusting for baseline Total Spitzer Quality of Life Index score, was assessed using the F-test from the ANCOVA. The model was as follows: Change in Total Spitzer Quality of Life Index Score = Baseline Total Spitzer Quality of Life Index Score + Treatment; Test type: Superiority or Other; p = 0.387, ANCOVA; Estimated mean treatment difference = 0.28, 95% CI 2-sided [-0.36 to 0.91]

7. Secondary Outcome: Patient Global Impression of Change at the End of 3 Weeks of Treatment.
Description: The Patient Global Impression of Change consisted of a single question relating to improvement in overall condition since the start of the study. The results were recorded as "Very Much Improved", "Much Improved", "Minimally Improved", "No Change", "Minimally Worse", "Much Worse" and "Very Much Worse" and were converted to a seven point scale ranging from one to seven, respectively. The number of patients who reported being "Very Much Improved" or "Much Improved" is presented.
Time Frame: 0 - 3 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 36 | 34
participants | 9 | 9
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The proportion of patients who considered their condition "Very Much Improved" or "Much Improved" was compared between treatment groups using a Fisher's Exact Test; Test type: Superiority or Other; p = 1.000, Fisher Exact; Estimated mean treatment difference = -1.47, 95% CI 2-sided [-21.56 to 18.51]

8. Secondary Outcome: Change From Baseline in Mean Pain Box Scale-11 Scores (Multiple Sclerosis Subset) at 3 Weeks.
Description: as for outcome 1
Time Frame: 0 - 3 weeks
Population: Patients whose entry into the study was as a result of pain related to Multiple Sclerosis were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 24 | 19
units on a scale | -1.6 (1.90) | -0.8 (1.60)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.128, ANCOVA; Estimated mean treatment difference = -0.86, 95% CI 2-sided [-1.97 to 0.26]

9. Secondary Outcome: Use of Analgesic Escape Medication - Multiple Sclerosis Subset.
Description: The percentage of days on treatment on which escape medication was used is presented.
Time Frame: 0 - 3 weeks
Population: Patients whose entry into the study was as a result of pain related to Multiple Sclerosis were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 24 | 19
percentage of days | 16.71 (28.55) | 48.48 (46.63)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; The proportions were compared between treatment groups using ANOVA with treatment as a factor; Test type: Superiority or Other; p = 0.009, ANOVA; Estimated mean treatment difference = -31.77, 95% CI 2-sided [-55.07 to -8.47]

10. Secondary Outcome: Change From Baseline in Mean Sleep Disturbance Scores (Multiple Sclerosis Subset) at 3 Weeks.
Description: as for outcome 3
Time Frame: 0 - 3 weeks
Population: Patients whose entry into the study was as a result of pain related to Multiple Sclerosis were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 24 | 19
units on a scale | -0.60 (0.89) | -0.36 (0.56)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.184, ANCOVA; Estimated mean treatment difference = -0.32, 95% CI 2-sided [-0.80 to 0.16]

11. Secondary Outcome: Change From Baseline in Mean Pain Disability Index Scores at 3 Weeks.
Description: as for outcome 4
Time Frame: 0 - 3 weeks
Population: Patients whose entry into the study was as a result of pain related to Multiple Sclerosis were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 17 | 16
units on a scale | -7.8 (11.26) | -1.7 (6.98)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.134, ANCOVA; Estimated mean treatment difference = -5.18, 95% CI 2-sided [-12.05 to 1.68]

12. Secondary Outcome: Change From Baseline in Mean Brief Pain Inventory (Short Form) Scores (Multiple Sclerosis Subset) at 3 Weeks.
Description: as for outcome 5
Time Frame: 0 - 3 weeks
Population: Patients whose entry into the study was as a result of pain related to Multiple Sclerosis were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 23 | 19
units on a scale | -4.5 (5.60) | -0.5 (5.06)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.031, ANCOVA; Estimated mean treatment difference = -3.77, 95% CI 2-sided [-7.17 to -0.36]

13. Secondary Outcome: Change From Baseline in Mean Spitzer Quality of Life Index Scores (Multiple Sclerosis Subset) at 3 Weeks.
Description: as for outcome 6
Time Frame: 0 - 3 weeks
Population: Patients whose entry into the study was as a result of pain related to Multiple Sclerosis were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 21 | 17
units on a scale | -0.1 (1.01) | 0.1 (1.64)
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.915, ANCOVA; Estimated mean treatment difference = 0.04, 95% CI 2-sided [-0.79 to 0.88]

14. Secondary Outcome: Patient Global Impression of Change - Multiple Sclerosis Subset.
Description: as for outcome 7
Time Frame: 0 - 3 weeks
Population: Patients whose entry into the study was as a result of pain related to Multiple Sclerosis were included in the analysis.
Measure: Number; unit: participants
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 24 | 19
participants | 6 | 4
Statistical Analysis 1: Comparison: GW-1000-02 vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 1.00, Fisher Exact; Estimated mean treatment difference = 3.95, 95% CI 2-sided [-21.85 to 27.47]

15. Secondary Outcome: Incidence of Adverse Events as a Measure of Patient Safety.
Description: The number of patients who experienced an adverse event in the study is presented.
Time Frame: 0 - 65 days
Population: All patients who entered the study, were randomised, received at least one dose of study medication and yielded on-treatment efficacy data were included in the safety analysis.
Measure: Number; unit: participants
Arm/Group | GW-1000-02 | Placebo
Number analyzed (Participants) | 36 | 34
participants | 35 | 26

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the time of consent to post study follow up (0 -5 weeks) were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | GW-1000-02 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/34
Other Adverse Events (participants affected / at risk) | 35/36 | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=36) | Placebo (N=34)
Sepsis Not Otherwise Specified (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=36) | Placebo (N=34)
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 2
Urinary Tract Infection Not Otherwise Specified (Infections and infestations) | 4 | 8
Dizziness (Nervous system disorders) | 20 | 5
Headache Not Otherwise Specified (Nervous system disorders) | 4 | 5
Gait Abnormal Not Otherwise Specified (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Dry Mouth (Gastrointestinal disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 2
Oral Discomfort (Gastrointestinal disorders) | 2 | 0
Oral Pain (Gastrointestinal disorders) | 2 | 2
Vomiting Not Otherwise Specified (Gastrointestinal disorders) | 2 | 0
Diarrhoea Not Otherwise Specified (Gastrointestinal disorders) | 0 | 3
Application Site Pain (General disorders) | 4 | 3
Fatigue (General disorders) | 4 | 0
Feeling Drunk (General disorders) | 3 | 0
Application Site Burning (General disorders) | 2 | 0
Feeling of Relaxation (General disorders) | 2 | 0
Lethargy (General disorders) | 2 | 0
Thirst (General disorders) | 2 | 0
Weakness (General disorders) | 2 | 0
Confusional State (Psychiatric disorders) | 3 | 0
Euphoric Mood (Psychiatric disorders) | 2 | 0
Paranoia (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 3
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Appetite Increased (Metabolism and nutrition disorders) | 3 | 0
Vision Blurred (Eye disorders) | 2 | 0
Pain in Limb (Musculoskeletal and connective tissue disorders) | 0 | 2
Back Pain Aggravated (Musculoskeletal and connective tissue disorders) | 0 | 2
Peripheral Swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Hypertension Not Otherwise Specified (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.